CLINICAL TRIAL: NCT01899079
Title: Prospective Observational Study to Evaluate the Impact of the Determination of the Intrinsic Subtypes of Breast Cancer by PAM50 NanoString Technology in the Use of Adjuvant Chemotherapy in Women With Breast Cancer, HR+ and Node -.
Brief Title: A Prospective Observational Study of Clinical Outcomes for the NanoString® Technologies Prosigna Gene Signature Assay
Status: Completed | Type: Observational
Sponsor: NanoString Technologies, Inc. (Industry)
Collaborators: Cedar Associates LLC (Other); Illumina, Inc. (Industry); Grupo Espanol de Investigacion del Cancer de Mama (Other); Spanish Breast Cancer Research Group (Other); Hospital General Universitario Gregorio Marañon (Other); Vall d'Hebron Institute of Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: PTL-00163
Record Dates: First submitted 2013-07-10; First posted 2013-07-15 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Prosigna; FFPE; node negative; estrogen receptor positive; HER2 negative
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — FFPE breast tumor tissue samples
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary objective of this study is to assess the extent to which the Prosigna™ Breast Cancer Prognostic Gene Signature Assay affects the medical oncologist's treatment recommendations regarding adjuvant chemotherapy and actual treatments received for patients with early-stage breast cancer.

DETAILED DESCRIPTION:
Changes in treatment recommendations will include (1) hormonal therapy alone, (2) hormonal therapy plus chemotherapy, and (3) changes in types of chemotherapy if chemotherapy was recommended before and after the Prosigna test.

ELIGIBILITY:
Inclusion Criteria:

* Resected node-negative, estrogen-receptor-positive, HER2-negative early- stage invasive breast cancer (T1-T2, N0, pN0 (i+), pN0 (mol+), M0)

  1. Estrogen receptor status will be evaluated by Immunohistochemistry (IHC)and more than 1% of stained tumor cells will be considered positive.
  2. HER2 status will be evaluated by (IHC; 0 or 1+, or 2+ will be considered negative) and by in-situ fluorescence hybridization.
* Postmenopausal females, which is defined as:

  1. Natural Amenorrhea > 12 months, regardless of age
  2. Bilateral oophorectomy, regardless of age (the oophorectomy must have been carried out at least 4 weeks before entering the study)
  3. Radiological castration with amenorrhea > 3 months, regardless of age
  4. Hysterectomy and postmenopausal blood levels
* Able to give consent
* Eligible for treatment of breast cancer with adjuvant chemotherapy
* ECOG performance status of 0 or 1

Exclusion Criteria:

* Tumor size T3-T4
* Non-invasive breast cancer (e.g., Paget's disease, DCIS)
* Tumors with nodes that are not N0, pN0 (i+), or pN0 (mol+)
* Tumors that are estrogen-receptor negative or HER2 positive
* Have metastatic disease
* Unable to give informed consent
* Unable to complete patient reported outcome surveys
* Have contraindications for adjuvant chemotherapy

  * Age, performance status, significant comorbidities
* ECOG performance status > 1

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Postmenopausal women with node-negative, estrogen-receptor positive, HER2-negative early-stage breast cancer. Investigators will offer enrollment to consecutively seen women who meet the entry criteria.
Sampling Method: Probability Sample
Enrollment: 217 (Actual)
Dates: Start 2013-06; Primary Completion 2014-01 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
The proportion of patients whose choice of treatment is changed as a result of receiving the Prosigna test result | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Martin, M.D., Ph.D., Principal Investigator — Hospital General Universitario Gregorio Marañón
Locations (7):
- Spain (7):
  - Consorci Sanitari de Terrassa, Barcelona
  - Corporacio Sanitaria Parc Tauli, Barcelona
  - Hospital U. Vall D'Hebron, Barcelona
  - Hospital U. Arnau de Vilanova, Lleida
  - Hospital G.U. Gregorio Maranon, Madrid
  - Hospital Quirón Madrid, Madrid
  - Hospital U. 12 de Octubre, Madrid